CLINICAL TRIAL: NCT00846872
Title: Effect of Continuous Subcutaneous GHRP-3 Infusion at 2 Dose Levels on the Physiological Secretion of the GH-IGF-I System, Blood Pressure, Glucose, Inflammatory Markers and Endothelial Function in Subjects With Insulin Resistance
Brief Title: Effect of Continuous GHRP-3 Infusion at on GH-IGF-I System, Blood Pressure, Glucose, and Insulin Resistance
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Inadequate subject recruitment
Sponsor: Tulane University Health Sciences Center (Other)
Responsible Party: Sponsor
Organization: Tulane University (Other)
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 65-08
Record Dates: First submitted 2009-02-17; First posted 2009-02-19 (Estimated); Last update posted 2021-01-08 (Actual); Status verified 2021-01

CONDITIONS: Insulin Resistance; Endothelial Dysfunction
Keywords: GHRP-3; Insulin Resistance; Markers of inflammation; Endothelial Dysfunction; Flow Mediated Dilation; GH/IGF-1 axis; Post menopausal
MeSH Terms: conditions — Insulin Resistance | interventions — Sodium Chloride; Mannitol

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Low dose GHRP-3 (Active Comparator): Subjects will receive the infusion for 14 ± 2 days. On day 1 of the test period, patients will report to the CTRC in a fasting state stay there for 3 - 4 hrs after the initiation of the infusion. Blood will be drawn in a fasting state and urine sample will be collected prior to insertion of the OmniPod and the CGMS. On day 7 +/- 2 days and on day 12 +/- 2 days, patients will report to the CTRC for blood draw and CGMS insertion. On day 14 +/- 2 days, patients will again report to CTRC for 24 hour admit. They will undergo urine sample collection, periodic blood draws and BP monitoring. After the 24 hour period, the CGMS will be disconnected and the patient will undergo FMD after which the test period will be terminated. There will be a washout period of 2 weeks between each test period.
  Interventions: Drug: GHRP-3 low dose
- High dose GHRP -3 (Active Comparator): Subjects will receive the infusion for 14 ± 2 days. On day 1 of the test period, patients will report to the CTRC in a fasting state stay there for 3 - 4 hrs after the initiation of the infusion. Blood will be drawn in a fasting state and urine sample will be collected prior to insertion of the OmniPod and the CGMS. On day 7 +/- 2 days and on day 12 +/- 2 days, patients will report to the CTRC for blood draw and CGMS insertion. On day 14 +/- 2 days, patients will again report to CTRC for 24 hour admit. They will undergo urine sample collection, periodic blood draws and BP monitoring. After the 24 hour period, the CGMS will be disconnected and the patient will undergo FMD after which the test period will be terminated. There will be a washout period of 2 weeks between each test period.
  Interventions: Drug: GHRP-3 high dose
- Saline Infusion (Placebo Comparator): Subjects will receive Placebo for 14 ± 2 days. On day 1 of the test period, patients will report to the CTRC in a fasting state stay there for 3 - 4 hrs after the initiation of the infusion. Blood will be drawn in a fasting state and urine sample will be collected prior to insertion of the OmniPod and the CGMS. On day 7 +/- 2 days and on day 12 +/- 2 days, patients will report to the CTRC for blood draw and CGMS insertion. On day 14 +/- 2 days, patients will again report to CTRC for 24 hour admit. They will undergo urine sample collection, periodic blood draws and BP monitoring. After the 24 hour period, the CGMS will be disconnected and the patient will undergo FMD after which the test period will be terminated. There will be a washout period of 2 weeks between each test period.
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: GHRP-3 low dose — 0.1 µg/kg/hr will be infused subcutaneously in a continuous manner using the Omnipod at the rate of 28 µl/hr
  Other Names: Formerly coded as 1485; Fourth generation growth hormone secretagogue
  Arms: Low dose GHRP-3
Drug: GHRP-3 high dose — 0.5 µg/kg/hr will be infused subcutaneously in a continuous manner using the Omnipod at the rate of 28 µl/hr
  Other Names: Formerly coded as 1485; Fourth generation growth hormone secretagogue
  Arms: High dose GHRP -3
Drug: Saline — 5% mannitol will be infused subcutaneously in a continuous manner using the Omnipod at the rate of 28 µl/hr
  Other Names: 5% mannitol
  Arms: Saline Infusion

SUMMARY:
The hypothesis is that GHRP-3 will exert beneficial effects on endothelial function and insulin resistance in older men and women via hormonal (GH, IGF-I, IGFBP-3,-1, insulin) and non-hormonal actions (anti-inflammatory).

DETAILED DESCRIPTION:
At the lower dose of 0.1 µg/kg/h, GHRP-3 presumably will improve endothelial dysfunction, enhance insulin action and lower blood pressure via the anti-inflammatory effects of GHRP-3 while at the higher dose of 0.5 µg/kg/h GHRP-3 these anti-inflammatory effects will be further augmented by the hormonal action of increasing serum IGF-I and its primary serum binding protein insulin like growth hormone binding protein - 3 (IGFBP-3 as well as -1). Also, the more detailed inter-relationships between the actions of GHRP-3, GH and IGF-I on serum glucose, blood pressure, and lipid levels over 24h periods will be determined at the end of the 14 day placebo and two GHRP-3 infusion periods. The GHRP-3 will be administered in escalating doses.

The Specific Aims of this study are as follows:

1. To determine the relative effects of 0.1µg/kg/h and 0.5µg/kg/h GHRP-3 as compared to placebo infusion in inducing physiological secretion of the GH-IGF-I system after continuous sc delivery for 14 days in healthy older men and women with insulin resistance.
2. To determine the relative interrelated effects of 0.1 and 0.5µg/kg/h GHRP-3 infusion and placebo on various hormonal and non hormonal aspects of insulin resistance such as blood pressure (BP), plasma glucose and FFA as well as GH, IGF-I, IGFBP-1, -3, insulin and endothelin-1 levels.
3. To determine the relative effects of placebo and the above 2 doses of GHRP-3 infusion on flow mediated dilation (FMD) and nitroglycerin-dependent dilation

ELIGIBILITY:
Inclusion Criteria:

1. Men and post-menopausal women 50-70 years.
2. Elevated fasting plasma glucose ranging <125 mg/dL
3. Waist circumference >35 inches in women and >40 inches in men

Exclusion Criteria:

1. Patients taking medications that may alter carbohydrate metabolism and/or insulin resistance.
2. Female patients with a positive pregnancy test.
3. Previous history of hypersensitivity to GHRP.
4. Patients with overt liver disease, renal disease and/or congestive heart failure.
5. Patients with anticipated change in medication regimen during the study period.
6. Current use or history of use of hormone replacement therapy in the last six months.
7. Current use or history of use of Ace Inhibitors or Angiotensin receptor blockers in the last six months.
8. Hemoglobin of < 11.6 g/dL for women and < 12.9 g/dL for men.

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-07; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Determine the relative effects of 0.1µg/kg/h and 0.5µg/kg/h GHRP-3 as compared to placebo in inducing physiological secretion of the GH-IGF-I system after continuous sc delivery in healthy older men and women with insulin resistance | 6 months

SECONDARY OUTCOMES:
Determine the relative interrelated effects of 0.1 and 0.5µg/kg/h GHRP-3 infusion and placebo on various hormonal and non hormonal aspects of insulin resistance. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Tina K Thethi, MD, MPH, Principal Investigator — AdventHealth